CLINICAL TRIAL: NCT03539081
Title: Investigating Mechanisms of Human Spinal Cord Stimulation for Purpose of Treating Restless Leg Syndrome
Brief Title: Spinal Cord Stimulation for Restless Legs Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marshall Holland (Other)
Responsible Party: Sponsor-Investigator, Marshall Holland, MD, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 201605777
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Restless Legs Syndrome; Neuropathic Pain
Keywords: Epidural Spinal Cord Stimulation; Muscle Sympathetic Nerve Activity; Blood Flow
MeSH Terms: conditions — Restless Legs Syndrome; Neuralgia | interventions — Absorptiometry, Photon; Blood Pressure Monitors; PO-2

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to one of two groups based on whether they have Restless Leg Syndrome to undergo experimental measurements that are made at each of the five measurement time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Subjects with RLS (Experimental): Subjects with Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  Interventions: Diagnostic Test: Dual-energy X-ray absorptiometry Scan; Other: Laboratory Measurements; Other: Blood Flow Measurement; Other: Partial pressure of oxygen; Other: Microneurography; Other: Anthropometric Measurements; Behavioral: John Hopkins Restless Legs Severity Scale
- Subjects without RLS (Other): Subjects without Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  Interventions: Diagnostic Test: Dual-energy X-ray absorptiometry Scan; Other: Laboratory Measurements; Other: Blood Flow Measurement; Other: Partial pressure of oxygen; Other: Microneurography; Other: Anthropometric Measurements
- Continous BP Monitoring (Other): This arm consists of subjects from arm "Subjects with RLS", "Subjects without RLS", and the rest of the qualifying subjects undergoing continuous blood pressure portion of the study only.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  Interventions: Other: Continuous Blood Pressure; Behavioral: Continuous Blood Pressure Diary

INTERVENTIONS:
Diagnostic Test: Dual-energy X-ray absorptiometry Scan — Body composition analysis will be obtained by DEXA scan.
  Other Names: DEXA
  Arms: Subjects with RLS; Subjects without RLS
Other: Laboratory Measurements — The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Arms: Subjects with RLS; Subjects without RLS
Other: Blood Flow Measurement — The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Arms: Subjects with RLS; Subjects without RLS
Other: Continuous Blood Pressure — Continuous Blood pressure cuff will worn for 2 days with spinal cord stimulator on and off (24 hour on and 24 hour off). Optional procedure.
  Other Names: 24-hour Ambulatory Blood Pressure Cuff
  Arms: Continous BP Monitoring
Other: Partial pressure of oxygen — Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Arms: Subjects with RLS; Subjects without RLS
Other: Microneurography — The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Arms: Subjects with RLS; Subjects without RLS
Other: Anthropometric Measurements — Height and weight will be obtained.
  Arms: Subjects with RLS; Subjects without RLS
Behavioral: John Hopkins Restless Legs Severity Scale — Subjects will be administered questionnaires to evaluate RLS symptoms using John Hopkins Restless Legs Severity Scale.
  Arms: Subjects with RLS
Behavioral: Continuous Blood Pressure Diary — Subjects participating in Continuous Blood Pressure monitoring will be administered continuous blood pressure monitoring compliance diary.
  Arms: Continous BP Monitoring

SUMMARY:
The overall goal of this proposed study is to evaluate the underlying mechanisms of neural control of blood flow in the lower extremities in humans with restless leg syndrome (RLS). At least 15% of the general public suffers from RLS and many more may go undiagnosed. This unfortunate disorder leads primarily to a disturbing sensation within the patient's lower extremities that requires movement for relief (1, 2). The central hypothesis of our study is that physiological changes in lower limb blood flow as a result of thoracolumbar epidural Spinal Cord Stimulation (SCS) lead to the relief of RLS.

DETAILED DESCRIPTION:
Patients age 18-85 years with (n=25) and without RLS (n=25) that have recently having undergone Spinal Cord Stimulation (SCS) implantation (thoracolumbar) for chronic pain will be recruited from the Departments of Anesthesia and Neurosurgery, University of Iowa Hospitals and Clinics. The rationale for studying both RLS patients and non-RLS patients with chronic back pain is to initially test the effectiveness of Spinal Cord Stimulation (SCS) on lower limb blood flow in the absence of symptoms of RLS. In the non-RLS patients, we could determine if SCS does in fact alter limb blood flow. We hypothesize that RLS patients have altered muscle sympathetic nerve activity (MSNA) and blood flow correlating to severity of RLS symptoms, which will then be modulated by Spinal Cord Stimulation (SCS), allowing for resolution of symptoms in RLS with MSNA-mediated improvements in leg blood flow. We also hypothesize that SCS in RLS patients will reduce 24-hour ambulatory blood pressure in parallel with reductions in MSNA.

Those deemed eligible to participate will be invited for 2 visits to the Translational Vascular Physiology Laboratory in the Clinical Research Unit (CRU) of the University of Iowa Hospitals and Clinics. Each of the 2 study visits are identical except for experimental measurements that are made at each of the five measurement time points when the Spinal Cord Stimulation (SCS) unit is either on or off as described below.

Visit 1: Experimental measurements include non-invasive "gold standard" measures of limb blood flow and arterial stiffness including femoral artery blood flow via Doppler ultrasound, calf blood flow from strain gauge venous occlusion plethysmography, and arterial stiffness via pulse wave velocity using applanation tonometry. Additionally, participants will be asked to assess the current level of leg discomfort every 10 minutes while measurements are taken by the SIT test, a validated technique for assessing restless legs symptoms where patients are asked to set and rest quietly during measurement talking, moving as little as possible (3).

Visit 2: Experimental measurements include direct measures of sympathetic nerve activity using microneurography before, during and again after administration of SCS to the patient. Additionally, participants will be asked to assess the current level of leg discomfort every 10 minutes while measurements are taken by the SIT test, a validated technique for assessing restless legs symptoms where patients are asked to set and rest quietly during measurement taking, moving as little as possible (3).

Some participates may visit the laboratory for placement of a 24-hour ambulatory blood pressure cuff.

ELIGIBILITY:
Inclusion Criteria:

* Mental capacity to understand and decide to participate in the research
* Recently have undergone or are planning to undergo SCS implantation (thoracolumbar region) for chronic pain.

Exclusion Criteria:

* Peripheral vascular disease
* History of ischemic heart disease ( examples myocardial infarction, cardiac bypass surgery, coronary stent, unstable angina)
* Heart transplantation
* Renal Failure
* Congestive heart failure
* Type 1 diabetes
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Holland, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohayon MM, O'Hara R, Vitiello MV. Epidemiology of restless legs syndrome: a synthesis of the literature. Sleep Med Rev. 2012 Aug;16(4):283-95. doi: 10.1016/j.smrv.2011.05.002. Epub 2011 Jul 26. PMID 21795081
- [Background] Earley CJ. Clinical practice. Restless legs syndrome. N Engl J Med. 2003 May 22;348(21):2103-9. doi: 10.1056/NEJMcp021288. No abstract available. PMID 12761367
- [Background] Garcia-Borreguero D, Kohnen R, Boothby L, Tzonova D, Larrosa O, Dunkl E. Validation of the Multiple Suggested Immobilization Test: A Test for the Assessment of Severity of Restless Legs Syndrome (Willis-Ekbom Disease). Sleep. 2013 Jul 1;36(7):1101-1109. doi: 10.5665/sleep.2820. PMID 23814348
- [Background] Cameron T. Safety and efficacy of spinal cord stimulation for the treatment of chronic pain: a 20-year literature review. J Neurosurg. 2004 Mar;100(3 Suppl Spine):254-67. doi: 10.3171/spi.2004.100.3.0254. PMID 15029914
- [Background] Foreman RD, Linderoth B. Neural mechanisms of spinal cord stimulation. Int Rev Neurobiol. 2012;107:87-119. doi: 10.1016/B978-0-12-404706-8.00006-1. PMID 23206679
- [Background] Yeh P, Walters AS, Tsuang JW. Restless legs syndrome: a comprehensive overview on its epidemiology, risk factors, and treatment. Sleep Breath. 2012 Dec;16(4):987-1007. doi: 10.1007/s11325-011-0606-x. Epub 2011 Oct 26. PMID 22038683
- [Background] Dauvilliers Y, Winkelmann J. Restless legs syndrome: update on pathogenesis. Curr Opin Pulm Med. 2013 Nov;19(6):594-600. doi: 10.1097/MCP.0b013e328365ab07. PMID 24048084
- [Background] Garcia-Borreguero D, Kohnen R, Silber MH, Winkelman JW, Earley CJ, Hogl B, Manconi M, Montplaisir J, Inoue Y, Allen RP. The long-term treatment of restless legs syndrome/Willis-Ekbom disease: evidence-based guidelines and clinical consensus best practice guidance: a report from the International Restless Legs Syndrome Study Group. Sleep Med. 2013 Jul;14(7):675-84. doi: 10.1016/j.sleep.2013.05.016. PMID 23859128
- [Background] Hornyak M, Scholz H, Kohnen R, Bengel J, Kassubek J, Trenkwalder C. What treatment works best for restless legs syndrome? Meta-analyses of dopaminergic and non-dopaminergic medications. Sleep Med Rev. 2014 Apr;18(2):153-64. doi: 10.1016/j.smrv.2013.03.004. Epub 2013 Jun 6. PMID 23746768
- [Background] Walters AS, Wagner ML, Hening WA, Grasing K, Mills R, Chokroverty S, Kavey N. Successful treatment of the idiopathic restless legs syndrome in a randomized double-blind trial of oxycodone versus placebo. Sleep. 1993 Jun;16(4):327-32. doi: 10.1093/sleep/16.4.327. PMID 8341893
- [Background] Goldberg LI. Dopamine receptors and hypertension. Physiologic and pharmacologic implications. Am J Med. 1984 Oct 5;77(4A):37-44. doi: 10.1016/s0002-9343(84)80036-4. PMID 6148892
- [Background] Wu M, Linderoth B, Foreman RD. Putative mechanisms behind effects of spinal cord stimulation on vascular diseases: a review of experimental studies. Auton Neurosci. 2008 Feb 29;138(1-2):9-23. doi: 10.1016/j.autneu.2007.11.001. PMID 18083639

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With RLS: Subjects with Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  First Visit (Day 1):
  Dual-energy X-ray absorptiometry Scan
  Laboratory Measurements: Pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg measured by ultrasonic probe on the skin over the femoral artery of leg and brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Anthropometric Measurements: Height and weight will be obtained.
  Visit 2 (Day 2):
  Laboratory Measurements repeated as done in Visit 1.
  Blood Flow Measurement repeated as done in Visit 1.
  Partial pressure of oxygen repeated as done in Visit 1.
  Microneurography: Sympathetic nervous system activity to subject's leg muscles measured by a tiny microelectrode placed in peroneal nerve in the leg located just below the outer knee. When the nerve is located 2 sterile microelectrodes will be inserted through the skin.
- Subjects Without RLS: Subjects without Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  First Visit (Day 1):
  Dual-energy X-ray absorptiometry Scan
  Laboratory Measurements: Pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg measured by ultrasonic probe on the skin over the femoral artery of leg and brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Anthropometric Measurements: Height and weight will be obtained.
  Visit 2 (Day 2):
  Laboratory Measurements repeated as done in Visit 1.
  Blood Flow Measurement repeated as done in Visit 1.
  Partial pressure of oxygen repeated as done in Visit 1.
  Microneurography: Sympathetic nervous system activity to subject's leg muscles measured by a tiny microelectrode placed in peroneal nerve in the leg located just below the outer knee. When the nerve is located 2 sterile microelectrodes will be inserted through the skin.
- Continous BP Monitoring: This arm consists of subjects from arm "Subjects with RLS", "Subjects without RLS", and the rest of the qualifying subjects undergoing continuous blood pressure portion of the study only.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  Continuous Blood Pressure: Continuous Blood pressure cuff will worn for 2 days with spinal cord stimulator on and off (24 hour on and 24 hour off). Optional procedure.
  Continuous Blood Pressure Diary: Subjects participating in Continuous Blood Pressure monitoring will be administered continuous blood pressure monitoring compliance diary.
Period: Overall Study
Arm/Group | Subjects With RLS | Subjects Without RLS | Continous BP Monitoring
Started | 5 | 10 | 0
Completed | 2 | 7 | 0
Not Completed | 3 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0
Not completed — MSNA testing not done due to nerve recording not being able to be done due to restless legs | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were no subjects enrolled in the Continuous BP Monitoring Arm
Groups:
- Subjects With RLS: Subjects with Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Intervention: Use of epidural spinal cord stimulation.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
  Continuous Blood Pressure Diary: Subjects participating in Continuous Blood Pressure monitoring will be administered continuous blood pressure monitoring compliance diary.
- Subjects Without RLS: Subjects without Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Intervention: Use of epidural spinal cord stimulation.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Continuous Blood Pressure: Continuous Blood pressure cuff will worn for 2 days with spinal cord stimulator on and off (24 hour on and 24 hour off). Optional procedure.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight
  John Hopkins Restless Legs Severity Scale
- Continous BP Monitoring: This arm consists of subjects from arm "Subjects with RLS", "Subjects without RLS", and the rest of the qualifying subjects undergoing continuous blood pressure portion of the study only.
  Intervention: Use of epidural spinal cord stimulation.
  Continuous Blood Pressure: Continuous Blood pressure cuff will worn for 2 days with spinal cord stimulator on and off (24 hour on and 24 hour off). Optional procedure.
  Continuous Blood Pressure Diary: Subjects participating in Continuous Blood Pressure monitoring will be administered continuous blood pressure monitoring compliance diary.
- Total: Total of all reporting groups
Arm/Group | Subjects With RLS | Subjects Without RLS | Continous BP Monitoring | Total
Number analyzed (Participants) | 5 | 10 | 0 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 4 | 10 |  | 14
  >=65 years | 1 | 0 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 7 |  | 9
  Male | 3 | 3 |  | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 1 | 0 |  | 1
  White | 4 | 10 |  | 14
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 10 |  | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change MSNA Burst Frequency From Baseline to 60 Minutes
Description: Response will measured by peroneal nerve microneurography to the lower limb during epidural spinal cord stimulation in patients with chronic back pain.
  Percent change MSNA burst frequency from baseline to 60 minutes
Time Frame: Baseline to 60 minutes
Population: All subjects enrolled did not complete this test or the test was terminated prior to a result being collected. The peroneal nerve signal is difficult to acquire and maintain with a small electrode through the skin, sometimes it can be lost half way if the patient moves their leg. Optional Continuous BP Monitoring did not have any subjects enrolled.
Measure: Mean (Standard Deviation); unit: Percent change MSNA burst frequency
Groups:
- Subjects With RLS: Subjects with Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
- Subjects Without RLS: Subjects without Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Subject will have received the standard of care intervention of epidural spinal cord stimulation for pain.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
  John Hopkins Restless Legs Severity Scale: Subjects will be administered questionnaires to evaluate RLS symptoms using John Hopkins Restless Legs Severity Scale.
Arm/Group | Subjects With RLS | Subjects Without RLS | Continous BP Monitoring
Number analyzed (Participants) | 1 | 4 | 0
Percent change MSNA burst frequency | -29 (1) | -24 (10) |

2. Primary Outcome: Response Measurement of Thoracolumbar Epidural SCS in the Femoral Artery Blood Flow
Description: The response will be measured by Doppler ultrasound of the femoral artery during epidural spinal cord stimulation in patients with chronic back pain.
Time Frame: Baseline and 1.5 Hours
Population: Not all subjects that were enrolled completed this test. Optional Continuous BP Monitoring sub-study did not have any participants enrolled.
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- Subjects With RLS: Subjects with Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Intervention: Use of epidural spinal cord stimulation.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
- Subjects Without RLS: Subjects without Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Intervention: Use of epidural spinal cord stimulation.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
  John Hopkins Restless Legs Severity Scale: Subjects will be administered questionnaires to evaluate RLS symptoms using John Hopkins Restless Legs Severity Scale.
Arm/Group | Subjects With RLS | Subjects Without RLS | Continous BP Monitoring
Number analyzed (Participants) | 4 | 8 | 0
percentage of change | 24 (30) | 22 (14) |

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events were collected during enrollment period, up to 2 months.
Description: Medical record review and directly from participants.
Groups:
- Subjects With RLS: Subjects with Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Intervention: Use of epidural spinal cord stimulation.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: The following labs will be obtained during the course of the study: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
  Continuous Blood Pressure Diary: Subjects participating in Continuous Blood Pressure monitoring will be administered continuous blood pressure monitoring compliance diary.
- Subjects Without RLS: Subjects without Restless Leg Syndrome that have recently undergone Spinal Cord Stimulation (SCS) Implantation for chronic pain.
  Intervention: Use of epidural spinal cord stimulation.
  Dual-energy X-ray absorptiometry Scan: Body composition analysis will be obtained by DEXA scan.
  Laboratory Measurements: pregnancy test (urine), glucose, insulin, catecholamine, and cholesterol (serum).
  Blood Flow Measurement: The blood flow to the arm or leg may also be measured by placing an ultrasonic probe on the skin over the femoral artery of the leg and the brachial artery of the arm.
  Partial pressure of oxygen: Transcutaneous recordings will be captured to measure the partial pressure of oxygen by placing monitors on the subject's chest and foot.
  Microneurography: The sympathetic nervous system activity to the subject's leg muscles will be measured by a tiny microelectrode placed in the peroneal nerve in the leg located just below the knee on the outer part of the leg. When the nerve is located 2 tiny sterile microelectrodes will be inserted through the skin.
  Anthropometric Measurements: Height and weight will be obtained.
  John Hopkins Restless Legs Severity Scale: Subjects will be administered questionnaires to evaluate RLS symptoms using John Hopkins Restless Legs Severity Scale.
  Continuous Blood Pressure Diary: Subjects participating in Continuous Blood Pressure monitoring will be administered continuous blood pressure monitoring compliance diary.
Arm/Group | Subjects With RLS | Subjects Without RLS | Continous BP Monitoring
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/10 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT03539081/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03539081/SAP_001.pdf
  • Informed Consent Form (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT03539081/ICF_002.pdf